CLINICAL TRIAL: NCT00411112
Title: Sentinel Node Study in Colon Cancer Surgery
Brief Title: Sentinel Node in Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3737
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Colon Cancer
Keywords: Sentinel node; Isosulphan blue; Isotopic detection; Survival
MeSH Terms: conditions — Colonic Neoplasms | interventions — RID

INTERVENTIONS:
Procedure: blue and isotopic detection of sentinel lymph nodes

SUMMARY:
More than 20% of patients operated on for colon cancer without node metastasis will develop visceral metastases. The purpose of the study is to determine sentinel lymph nodes with two methods: blue injection and isotopic detection. Sentinel nodes will then be analyzed by immunohistochemy to detect micrometastases. No adjuvant therapy will be proposed to the patient if there are only node's micrometastases and survival will be analyzed in regard to the presence of these micrometastasis.

ELIGIBILITY:
Inclusion Criteria:

* adult
* colon cancer
* open surgery

Exclusion Criteria:

* emergency surgery
* metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2007-03; Primary Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Survival without recurrence after 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Brigand, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Générale et Digestive - Hôpital de Hautepierre, Strasbourg, France